CLINICAL TRIAL: NCT03163316
Title: The Role of Unenhanced Magnetic Resonance Imaging in Quantitative Assessment of Metastatic Involvement of Axillary Lymph Nodes in Patients With Breast Cancer: Observational Descriptive Study.
Brief Title: The Role of Magnetic Resonance Imaging in Assessment of Axillary Lymph Nodes Metastasis in Breast Cancer Patients.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sandy Harby, Principal Investigator, Assiut University
Other Study IDs: MRIALBC
Record Dates: First submitted 2017-05-20; First posted 2017-05-23 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients: Patients will undergo unenhanced magnetic resonance imaging on both axillae.
  Interventions: Other: Unenhanced magnetic resonance imaging.

INTERVENTIONS:
Other: Unenhanced magnetic resonance imaging. — The axillary lymph nodes will be evaluated on axial Time 1-weighted images obtained without fat saturation. We will measure the largest dimension and cortical thickness of each lymph node and ratio of the two measurements will be calculated.
  The lymph nodes seen in Time 1-weighted images will be subsequently identified on the diffusion-weighted images to calculate the apparent diffusion coefficient value of each lymph node.
  Axillary lymph nodes scanned by magnetic resonance imaging will be compared by results of histopathological examination.

SUMMARY:
Breast cancer is the most common cancer among women worldwide.The main cause of cancer related death is the invasion and metastasis. The usual site of spread outside the breast is to lymph nodes in the axilla.

DETAILED DESCRIPTION:
The presence of axillary metastasis is important for prognosis and determining of treatment plan, so identification of axillary metastasis in early stage newly diagnosed breast cancer is important for staging of disease and treatment. However, approximately 40% of women who presents with early stage breast cancer also have axillary metastasis.

The status of lymph nodes in patients with breast cancer used to be evaluated with axillary lymph node dissection. During the last 15 years, sentinel lymph node biopsy has replaced for grading of patients with clinically lymph node negative breast cancer. Despite being a less invasive method when compared to axillary lymph node dissection, sentinel lymph node biopsy also leads to complications such as lymphedema, seroma, localized swelling, pain, paresthesia, decrease in arm strength, infectious neuropathy and shoulder stiffness in 20% of patients.

The imaging modalities for assessing the axillary lymph nodes are rapidly evolving. Ultrasound is applied widely for its convincing and dynamic observation. However, the sensitivity and specificity of ultrasound for lymph node metastasis were unreliable and controversial.

Owing to radiation and relative lower diagnostic accuracy, computed tomography is limited in clinic.

Positron emission tomography and positron emission tomography/computed tomography can reflect metabolism of glycolytic activity. Undoubtedly, they have shown the higher diagnostic significance in assessing distant metastasis and regional metastatic axillary lymph nodes, but their high radiation and expensive fee keep the common people away. Ultrasmall super paramagnetic iron oxide is the same.

Magnetic resonance imaging is developing with an unimaginable speed. Over the past years, it has been used to evaluate axillary lymph nodes. Its sensitivity and specificity for metastatic axillary lymph nodes were higher than ultrasound and computed tomography.

Diffusion weighted imaging is an advanced magnetic resonance imaging application which derives its image contrast from the differences in water mobility in the extracellular spaces, reflecting cellular density, organization, microstructure and microcirculation.

Several studies have shown that diffusion weighted imaging can serve as a powerful tool for differentiating benign from malignant breast lesions. In addition to this use, diffusion weighted imaging may also be used in the assessment of axillary lymph nodes, since they show similar tissue characteristics to the primary tumor.

Evaluation of lymph nodes is a promising novel application of diffusion weighted imaging , which can easily be applied as an adjunct to conventional breast magnetic resonance imaging . There are a few preliminary studies that have shown that diffusion weighted imaging can be used to detect lymph nodes affected by malignant cells. Koh reported that after the involvement of nodes with malignancy, they undergo changes and the increase in cellularity leads to diffusion restriction and low apparent diffusion coefficient values.

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients who proved positive for primary breast cancer by histopathology with axillary lymph nodes detected clinically or with superficial ultrasound on both axillae.

2) The included lymph nodes with minimal axial diameter (4mm).

Exclusion Criteria:

* 1)Patients who have a heart pacemaker as they are absolutely contraindicated for magnetic resonance imaging.

  2) Patients with severe claustrophobia. 3) Patients undergoing any type of neoadjuvant chemo-, immune- or endocrine therapy.

  4) Patients with history of axillary surgery or treatment. 5) Patients with recurrent axillary disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients who are coming to South Egypt Cancer Institute- Assiut University and proved positive for primary breast cancer by histopathology with axillary lymph nodes detected clinically or with superficial ultrasound on both axillae.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of unenhanced magnetic resonance imaging in assessment of axillary lymph node metastasis in breast cancer patients. | one month
  number of malignant axillary lymph nodes are accurately diagnosed by unenhanced magnetic resonance imaging in compared with histopathological result.

CONTACTS AND LOCATIONS:
Overall Officials: Sandy HN Ghaly, MBBCh, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Asyut
  - South Egypt Cancer Institute, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harnan SE, Cooper KL, Meng Y, Ward SE, Fitzgerald P, Papaioannou D, Ingram C, Lorenz E, Wilkinson ID, Wyld L. Magnetic resonance for assessment of axillary lymph node status in early breast cancer: a systematic review and meta-analysis. Eur J Surg Oncol. 2011 Nov;37(11):928-36. doi: 10.1016/j.ejso.2011.07.007. Epub 2011 Aug 19. PMID 21855267
- [Background] Heusner TA, Kuemmel S, Hahn S, Koeninger A, Otterbach F, Hamami ME, Kimmig KR, Forsting M, Bockisch A, Antoch G, Stahl A. Diagnostic value of full-dose FDG PET/CT for axillary lymph node staging in breast cancer patients. Eur J Nucl Med Mol Imaging. 2009 Oct;36(10):1543-50. doi: 10.1007/s00259-009-1145-6. Epub 2009 May 5. PMID 19415270
- [Background] Harada T, Tanigawa N, Matsuki M, Nohara T, Narabayashi I. Evaluation of lymph node metastases of breast cancer using ultrasmall superparamagnetic iron oxide-enhanced magnetic resonance imaging. Eur J Radiol. 2007 Sep;63(3):401-7. doi: 10.1016/j.ejrad.2007.02.010. Epub 2007 Mar 29. PMID 17398053
- [Background] Bedi DG, Krishnamurthy R, Krishnamurthy S, Edeiken BS, Le-Petross H, Fornage BD, Bassett RL Jr, Hunt KK. Cortical morphologic features of axillary lymph nodes as a predictor of metastasis in breast cancer: in vitro sonographic study. AJR Am J Roentgenol. 2008 Sep;191(3):646-52. doi: 10.2214/AJR.07.2460. PMID 18716089
- [Background] Koh DM, Collins DJ. Diffusion-weighted MRI in the body: applications and challenges in oncology. AJR Am J Roentgenol. 2007 Jun;188(6):1622-35. doi: 10.2214/AJR.06.1403. PMID 17515386